CLINICAL TRIAL: NCT00513630
Title: Phase 4 Study on the Prognosis and Effect of Anti-diabetic Drugs on Type-2 Diabetes Mellitus With Coronary Artery Disease
Brief Title: Study on the Prognosis and Effect of Anti-diabetic Drugs on Type-2 Diabetes Mellitus With Coronary Artery Disease
Acronym: SPREADDIMCAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCEMD002
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2010-12

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Glipizide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Active Comparator)
  Interventions: Drug: Glipizide
- glipizide (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Glipizide
  Arms: metformin
Drug: Metformin
  Arms: glipizide

SUMMARY:
The purpose of this study is to explore the recurrence risk of cardiovascular events in patients with type 2 diabetes mellitus and coronary heart disease after different antidiabetic drug therapy (glipizide or metformin) by using an double-blind, randomized, parallel control and prospective study

The end point of this study is:

1. follow up 3yr
2. recurrence of cardiovascular event
3. death caused by other reasons such as stroke, uremia, blindness and amputation

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease
* Type 2 diabetes

Exclusion Criteria:

* Severe organ dysfunction, psychopathy, infection, neutropenia
* Congenital heart disease, rheumatic heart disease, severe arrhythmia, myocardiopathy

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2004-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Composite of cardiovascular events which were defined as death from a cardiovascular cause, death from any cause, nonfatal myocardial infarction, nonfatal stroke or arterial revascularization

SECONDARY OUTCOMES:
New or worsening angina
new or worsening heart failure
new critical cardiac arrhythmia
new peripheral vascular events

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD. PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Hong J, Zhang Y, Lai S, Lv A, Su Q, Dong Y, Zhou Z, Tang W, Zhao J, Cui L, Zou D, Wang D, Li H, Liu C, Wu G, Shen J, Zhu D, Wang W, Shen W, Ning G; SPREAD-DIMCAD Investigators. Effects of metformin versus glipizide on cardiovascular outcomes in patients with type 2 diabetes and coronary artery disease. Diabetes Care. 2013 May;36(5):1304-11. doi: 10.2337/dc12-0719. Epub 2012 Dec 10. PMID 23230096